CLINICAL TRIAL: NCT01766609
Title: Efficacy and Safety of Intralesional Triamcinolone Acetonide in Vitiligo: A Prospective, Double-Blind Randomized Controlled Trial
Brief Title: Efficacy and Safety of Intralesional Corticosterois in the Treatment of Vitiligo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H12-02140
Record Dates: First submitted 2013-01-09; First posted 2013-01-11 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Vitiligo
Keywords: Vitiligo; Intralesional; Triamcinolone acetonide
MeSH Terms: conditions — Vitiligo | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Triamcinolone acetonide (Active Comparator): Injections will be given within one half of a single vitiligo patch. The concentration of triamcinolone acetonide (TA) that will be used initially is 2.5 mg/ml. Dilution will be done using a bacteriostatic normal saline. Each half will receive injections with either TA 2.5 mg/ml or normal saline as a control. Only one investigator will know the intervention each half has received. If the patient did not show any evidence of repigmentation during the 3rd visit (i.e. after two injection sessions with TA 2.5 mg/ml) , the concentration of TA will be increased to 5 mg/ml. A total of 4 injections will be given over 4 visits. The treatment will be repeated every 3 to 5 weeks for a total of 4 treatment sessions.
  Interventions: Drug: Triamcinolone Acetonide
- B: Normal saline (Placebo Comparator): Bacteriostatic normal saline will injected into one half of the vitiligo patch.

INTERVENTIONS:
Drug: Triamcinolone Acetonide
  Arms: A: Triamcinolone acetonide

SUMMARY:
Vitiligo is a chronic acquired disease characterized by well defined white macules and patches affecting the skin. It has a major psychosocial impact on affected patients. There are many treatment modalities available for vitiligo, however, none of them cure the disease. Topical corticosteroids (CS) are the most effective monotherapy for localized vitiligo. Treatment with intralesional corticosteroids (ILCS) is commonly used in many dermatologic conditions. However, there are only a few studies published on the use of ILCS in vitiligo. This is a prospective double-blind randomized clinical trial to assess efficacy and safety of ILCS in the treatment of vitiligo. Four treatment sessions will be done over 4 to 6 months. The investigators will compare intralesional triamcinolone acetonide (active treatment) to normal saline (placebo).

DETAILED DESCRIPTION:
Vitiligo is a chronic acquired disease characterized by well defined white macules and patches affecting the skin and mucous membranes. Mucocutaneous lesions develop secondary to selective destruction of melanocytes. It has a major psychosocial impact on affected patients. The etiology of vitiligo is largely unknown but more likely to be multifactorial. There are several theories on the pathogenesis of vitiligo including mainly the autoimmune, neurohormonal, and autocytotoxic theories. The autoimmune hypothesis has the strongest evidence with alteration mainly in the cellular immune response.

Diagnosis of vitiligo is usually made clinically. A skin biopsy is rarely needed for diagnosis and typically shows absence of melanin in the epidermis with no or few melanocytes. Perivascular inflammation has been found in approximately 92% of cases. Spontaneous repigmentation is uncommon (seen in 10-20% of patients) in vitiliginous patches but can occur. Repigmentation occurs usually in a perifollicular pattern, suggesting that the hair follicle functions as a reservoir for melanocytes.

There are many treatment modalities available for vitiligo, however, none of them cure the disease. These include different topical treatments, phototherapy, surgical therapy, and depigmentation therapy. Topical corticosteroids (CS) are commonly used as a first-line therapy for localized vitiligo. They are the most effective monotherapy for localized vitiligo. Studies have shown an increase in inflammatory cells in vitiliginous skin, mainly macrophages and T cells. Efficacy of CS in vitiligo is attributed to modulation of the immune response, reduction of destruction of melanocytes, and induction of melanocyte proliferation and melanin production. Treatment with intralesional corticosteroids (ILCS) is commonly used in many dermatologic conditions. There are only a few studies published on the use of ILCS in vitiligo. Triamcinolone acetonide (TA) is the most commonly used form of ILCSs. It is characterized by low solubility, being slowly absorbed from the injection site, prompting maximal local action, limiting diffusion and spread through tissue, and not giving rise to systemic side effects if used in therapeutic doses. The concentration that is most commonly used in dermatology is 2.5 mg/ml.

Side effects of intralesional TA (IL TA) include pain at the injection site, mild bleeding, transient atrophy and telangiectasia, hypopigmentation, and hyperpigmentation. Infection is uncommon but caution over bony prominences is recommended. It has been shown that TA at a total dose of 20 mg does not result in adrenal suppression. Hypersensitivity reactions to TA or the vehicle carboxymethylcellulose are extremely rare.

The investigators' hypothesis is that IL TA will induce significant skin pigmentation to improve vitiligo. This due to the anti-inflammatory effect of IL TA. IL TA has been successfully used in the treatment of many skin conditions with an autoimmune pathogenesis including alopecia areata. The investigators plan on conducting a prospective double-blind randomized clinical trial to assess efficacy and safety of IL TA in the treatment of vitiligo.

Study Objectives

1. To evaluate the potential for IL TA to induce repigmentation within vitiligo patches.
2. To assess the side effect profile of IL TA when used in the treatment of vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Localized or generalized vitiligo that involves a non mucosal or acral site.
* Patients should have a patch of at least 5 cm in the smallest diameter that shows no more than 10% repigmentation as assessed visually

Exclusion Criteria:

* Patients who received treatment for vitiligo within the past 4 weeks.
* Hypersensitivity to TA or vehicle.
* Pregnancy or breast-feeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-10 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the degree of repigmentation based on the modified VASI score for each half. We will consider the treatment successful if there was ≥50% change in modified VASI score from baseline. | 3-5 weeks after each treatment session

SECONDARY OUTCOMES:
Assessment of side effects in each half including atrophy, telangiectasia, hyperpigmentation and hypopigmentation using a severity scale as follows: 0=none, 1=mild, 2=moderate, 3=severe. | 3-5 weeks after each treatment session

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Lui, MD, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- The Skin Care Center, Vancouver General Hospital, Vancouver, British Columbia, Canada